CLINICAL TRIAL: NCT00526721
Title: An Observational, Non-interventional, Multi-center Study to Evaluate Efficacy and Tolerability of High Dose Rosuvastatin in High Risk Patients After Titration
Brief Title: Real-life EValuation Of High Dose RosUvastatin in High Risk Patients After TitraTION
Acronym: REVORUTION
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CKR-CRE-2007/6
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia; Crestor; LDL target goal; high risk patients; Naturalistic; Observational
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate achievement ratio of treatment target goal in hypercholesterolemia patients with high risk after high dose rosuvastatin(20mg/day) titration

ELIGIBILITY:
Inclusion Criteria:

* High-risk hyperlipidemia patients who are prescribed with rosuvastatin 10mg, based on the physician's clinical decision and fulfill the following criteria

  1. Over 18 years of age
  2. Have history of CHD or CHD risk equivalents, such as peripheral arterial disease, abdominal aortic aneurysm, symptomatic carotid artery disease (TIA or stroke of carotid origin or >50% obstruction of carotid artery), DM, and 2+ risk factors with 10-year risk CHD>20%

Exclusion Criteria:

1. Patients already taking other hyperlipidemic agents
2. Patients who do not fulfil the indication criteria for statin therapy
3. Patients who do not have baseline and/or follow-up lipid data to verify the efficacy data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypercholesteromia patients with high risk according to NCEP ATP III guideline in Korean tertiary care centers
Sampling Method: Probability Sample
Enrollment: 1482 (Actual)
Dates: Start 2007-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyunah Caroline Choi, Study Director — AstraZeneca Korea
Locations (3):
- South Korea (3):
  - Research Site, Seoul, Jongro-gu
  - Research Site, Seoul, Kangnam-gu
  - Research Site, Seoul, Songpa-gu